CLINICAL TRIAL: NCT02985229
Title: Acceptability and Feasibility of Medical Abortion in Singapore: A Study of 800 μg Buccal Misoprostol Following 200 mg Mifepristone for Abortion Through 70 Days Gestation
Brief Title: Acceptability and Feasibility of Medical Abortion in Singapore
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1028
Record Dates: First submitted 2016-10-19; First posted 2016-12-07 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Medical Abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Experimental): All participants in the study will be given the option of home administration of 200 mg oral mifepristone and 800 μg buccal misoprostol for medical abortion.
  Interventions: Drug: Mifepristone; Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — The option of home or clinic administration of 200 mg oral mifepristone
Drug: Misoprostol — 800 μg buccal misoprostol through 70 days LMP following administration of mifepristone

SUMMARY:
To test the hypothesis that a regimen of 200 mg oral mifepristone, with the option of home administration, followed by 800 μg buccal misoprostol 24 hours later for abortion through 70 days LMP will be feasible and acceptable in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* Have an intrauterine pregnancy consistent wit gestational age ≤ 70 days
* Be 21 years of age or over
* Be willing and able to sign consent forms
* Be eligible for abortion according to current hospital guidelines
* Be able to return to the clinic and able to contact study staff or emergency medical services if needed
* Be willing to provide an address, email and/or telephone number for purposes of follow-up
* Agree to comply with the study procedures and visit schedule

Exclusion Criteria:

* confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass
* chronic renal failure
* concurrent long-term corticosteroid therapy
* history of inherited porphyrias
* IUD in place (must be removed after mifepristone is administered).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Rate of successful abortion | 7-10 days after mifepristone administration
  Proportion of abortions that are complete without surgical intervention

SECONDARY OUTCOMES:
Satisfaction with the medical abortion method | 7-10 days after mifepristone administration
  Proportion of women who are satisfied with the medical abortion method
Preferred location of mifepristone administration | The day of enrollment
  Proportion of women who select home use of mifepristone

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (2):
- Singapore (2):
  - KK Women's and Children's Hospital, Singapore
  - National University Hospital, Singapore